CLINICAL TRIAL: NCT05677412
Title: Sleep, Pain and Stress in Adolescents With Persistent Pain
Acronym: PedPainSleep
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Helsinki University Central Hospital (Other)
Collaborators: University of Helsinki (Other)
Responsible Party: Principal Investigator, Reetta Sipilä, Head of research, Helsinki University Central Hospital
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Treatment
Other Study IDs: ULSHelsinki
Record Dates: First submitted 2023-01-03; First posted 2023-01-10 (Actual); Last update posted 2025-09-15 (Actual); Status verified 2025-09

CONDITIONS: Pain, Chronic; Sleep
MeSH Terms: conditions — Chronic Pain

STUDY DESIGN:
Intervention Model Description: Experimental within-subject study design
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- neutral story (Active Comparator): Neutral story before the sleep onset
  Interventions: Behavioral: Neutral story
- suggestive story (Experimental): Suggestive story to find out the effect of relaxation to sleep structures.
  Interventions: Behavioral: suggestive relaxation

INTERVENTIONS:
Behavioral: suggestive relaxation — suggestive story before sleep onset
  Arms: suggestive story
Behavioral: Neutral story — neutral story before sleep
  Arms: neutral story

SUMMARY:
The main aim is the gain information of sleep structures in adolescents with persistent pain. Also to study simple interventions to support their sleep and pain management. The main aim of this study is to test the efficacy and feasibility of suggestive presleep relaxation technique in improving sleep quality and sleep-related emotional memory processing.

ELIGIBILITY:
Inclusion Criteria:

* Patients aged 15-17 years with persistent (> 3months) pain reporting average pain intensity over 3/10 on the Numerical Rating Scale (NRS).

Exclusion Criteria:

* ongoing medication for sleep or pain.

Ages: 15 Years to 17 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 20 (Estimated)
Dates: Start 2023-05-23 (Actual); Primary Completion 2026-06-30 (Estimated); Study Completion 2026-06-30 (Estimated)

PRIMARY OUTCOMES:
Sleep quality | one night
  The overnight PSG (Somnomedics) is used to measure sleep during two nights (Somnomedics, Somnoscreen plus HD), with the following recorded parameters: electroencephalography (left and right for F, C, O); left and right eletrooculogram; left and right electromyogram; electrocardiogram. Sleep recordings are done with portable devices so that the patients will sleep at their home during the recordings.

CONTACTS AND LOCATIONS:
Locations (1):
- New Childrens Hospital, Helsinki, Finland

IPD SHARING:
Plan to Share IPD: No